CLINICAL TRIAL: NCT04295083
Title: The Effect of Clay Based Group Study on the Loneliness and Hopelesness Levels in Elderly Living Alone: Randomized Controlled Study
Brief Title: Effect of Clay Based Group Study With Elderly Living Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Merve Aydın, Principal Investigator, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nurse_Psychiatric61
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: ART
Keywords: clay therapy; psychiatric nurse; loneliness; hopelessness; elderly

STUDY DESIGN:
Who Masked: Participant
Masking Description: Without knowing that participants are in the experimental or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will be six 1,5 h weekly of clay based group study and interviewed face-to-face twice by the researchers.
  Interventions: Behavioral: clay based group study
- Control group (No Intervention): The control group will interviewed face-to-face twice

INTERVENTIONS:
Behavioral: clay based group study — Clay based group work sessions were applied to the experimental group for 60-90 minutes once a week for 6 weeks. The sessions are composed of structured or semi-structured activities prepared for the purpose of the literature by the researcher for the purposes such as acquiring new solutions and life skills to reduce loneliness and hopelessness of individuals aged 65 and over, and sharing their feelings, thoughts, and memories with other individuals. Clay Study Activity Booklet ". Four expert opinions were obtained for the booklet created. Methods such as narration, sharing experiences, group practice, question-answer, learning by doing, imagining were used in the activity program. The physical, psychological, social and mental characteristics of the elderly were taken into consideration in the selection of these methods.
  Arms: Experimental group

SUMMARY:
This study determines the effectiveness of clay-based group study on the loneliness and hopelessness levels in elderly living alone. For this, while the experimental group will six 1,5 h weekly of clay-based group study and interviewed face-to-face twice, the control group will interview face-to-face twice

DETAILED DESCRIPTION:
One of the most important social changes today is the aging of the world's population. Along with the increasing elderly population, there is a serious increase in the number of elderly living alone. Many problems such as living alone, despair, insecurity, fear, depression, future anxiety, and close relationship longing are seen in the elderly who constitute the risk group in terms of mental health. The communication, social life and support opportunities of the elderly living alone with other people, their environment, relatives, and society are decreasing. Today, loneliness is one of the most commonly experienced psychological symptoms among the elderly. It has been reported that the feeling of loneliness is 80.0% in individuals aged 65 and over, and the age when this feeling is most common is 70 and above. Another of the most common emotions in the elderly is hopelessness. It is recommended to use art therapy, which is a supportive method suitable for a biopsychosocial approach in coping with loneliness and hopelessness. The art type, technique, and materials to be used in art therapy should be compatible with the age, ability, mental and physical development of the person to be applied. It is a substance that can be manipulated and deformed many times due to its clay structure. The person doing the clay works without fear of damaging the object due to the plastic and durable structure of the clay. Due to its advantage of being able to do it comfortably, it is a suitable art form for elderly individuals who are in the period of neurocognitive decline. Under this scope, this study will evaluate the effect of clay-based group study on the loneliness and hopelessness levels in elderly living alone.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years and old,
* To get a score of 19 and above on the Mini-Mental Status examination scale,
* Scoring less than 30 on the Beck Depression scale,
* To score 32 and above on UCLA-LS Loneliness scale,
* To get 4 points or more from the Beck Hopelessness Scale,
* Volunteering to participate in the research

Exclusion Criteria:

* Having a perception disorder that will prevent communication,
* Having a neurological and physical discomfort (paralysis, rheumatoid arthritis, etc.) in their hands,
* Having been diagnosed with any mental disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — 65 Years and older
Enrollment: 60 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Measurement of Loneliness | 6 weeks
  At the end of 6 weeks (6 sessions of clay work + 2 sessions face to face interview), they will be evaluated using the UCLA-LS Loneliness Scale. The highest score that can be obtained from the scale is 80, and the lowest score is 20. High scores show that individuals experience more loneliness. 20-31 score range "No loneliness", 32-41 score range "Very mild loneliness", 42-53 score range "Slight loneliness", 54-67 score range "Lonely" and 68-80 score range is classified as "Totally lonely". The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Measurement of Hopelessness | 6 weeks
  At the end of 6 weeks (6 sessions of clay work + 2 sessions face to face interviews) will be evaluated using the Beck Hopelessness Scale. The highest score that can be obtained from the scale is 20, and the lowest score is 1. When the scores are high, the hopelessness of the individual is assumed to be high. 0-3 points of hopelessness, 4-8 points of low hopelessness, 9-14 points of medium hopelessness and 15-20 points of high hopelessness were stated. It is stated that it can be used to predict suicide for scores of 9 and above. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: merve aydın, Principal Investigator — Karadeniz Technical University
Locations (2):
- Turkey (Türkiye) (2):
  - Merve Aydın, Trabzon, Karadeniz Technical University
  - Yasemin Kutlu, Istanbul

IPD SHARING:
Plan to Share IPD: No
There is no plan to share to IPD

REFERENCES:
- [Derived] Aydin M, Kutlu FY. The Effect of Group Art Therapy on Loneliness and Hopelessness Levels of Older Adults Living Alone: A Randomized Controlled Study. Florence Nightingale J Nurs. 2021 Oct;29(3):271-284. doi: 10.5152/FNJN.2021.20224. PMID 35110167